CLINICAL TRIAL: NCT00005206
Title: Calcium Intake, Metabolism, and Gestational Blood Pressure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1085; R01HL040005 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To determine if low dietary calcium intake and disturbances in maternal calcium metabolism were associated with increases in blood pressure in late pregnancy.

DETAILED DESCRIPTION:
BACKGROUND:

The importance of maintaining dietary calcium intake and normal calcium metabolism for optimal regulation of arterial blood pressure has been demonstrated in humans and animals. Recent reports have suggested that low dietary calcium intake and disturbances in maternal calcium metabolism are associated with increases in blood pressure in late gestation. These factors may be associated with an increased risk of developing pregnancy-induced hypertension.

This study was conducted in response to a Request for Applications on Research on Hypertension in Pregnancy jointly released in 1986 by the National Heart, Lung, and Blood Institute and the National Institute of Child Health and Human Development.

DESIGN NARRATIVE:

Blood pressure, nutrient intake, and markers of calcium metabolism were prospectively assessed in normal, pregnant women. Nutrient intakes, including dietary calcium, were assessed during gestation weeks 24, 28, 32, 36, and the postpartum period using 3-day food records and 24-hour dietary recalls. Concomitantly, serum measures of calcium metabolism were assessed including serum total and ionized calcium, parathyroid hormone, calcitonin, vitamin D concentration, serum magnesium, phosphorus, sodium, and potassium concentrations. During weeks 24 and 32, urinary excretion of sodium, calcium, magnesium, potassium, phosphorus, cAMP, and creatinine were measured. Blood pressures were measured at every prenatal visit and postpartum. Measures of infant growth and blood pressure were assessed at 1, 6, and 12 months of age to determine if maternal dietary calcium intake exerted long-term influences on infant development and blood pressure.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-09; Study Completion 1991-08 (Actual)